CLINICAL TRIAL: NCT06450080
Title: Study of the Relationship Between Clinical, Imaging and Biological Data in Patients With Squamous Cell Carcinoma of the Tongue
Acronym: ClimaBio
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PI2024_843_0036
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Soft Tissue Tumors of the Tongue; Squamous Cell Carcinoma; Proton Magnetic Resonance Spectroscopy; Transcriptomics
Keywords: Tongue tissue; Squamous Cell Carcinoma; proton magnetic resonance spectroscopy; 1H-MRS; spectroscopic and metabolic profile; noninvasive biomarkers; Transcriptomics
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients (Experimental): Patients with a lingual tumor measuring less than 15 mm in long axis
  Interventions: Other: MRI and MRS acquisitions
- healthy volunteers (Active Comparator): Subjects without a history of cancer of the upper aerodigestive tract Subjects without contraindication to MRI Subjects over 18 years old Subjects who have provided free and informed written consent Subjects benefiting from a social security system
  Interventions: Other: MRI and MRS acquisitions

INTERVENTIONS:
Other: MRI and MRS acquisitions — All MRI and MRS acquisitions for this study will be carried out on the GIE Faire Faces ACHIEVA 3T TX DStream Philips® Research MRI using a 32-channel head antenna located at the Amiens-Picardie University Hospital .

SUMMARY:
Squamous cell carcinoma (SCC) could be a very aggressive cancer and has a bad prognosis if not detected early and thus is associated with high mortality. The development of simple and reliable biomarkers for the early detection of SCC is one of the solutions to better diagnose, treat these tumors, evaluate and monitor treatments, and hence reduce mortality. In a previous work, the investigators demonstrated the ability of Proton Magnetic resonance spectroscopy (1H-MRS) to non-invasively assess spectroscopic and metabolic profiles of tongue tissue in healthy subjects. In the present work, the investigators challenge the use of in-vivo 1H-MRS as a potential method for non-invasive metabolic monitoring of patients with squamous cell carcinoma of the tongue undergoing therapy. Thus the main objective is to study the spectroscopic and metabolic differences, e.g. including variation in the metabolite TMA-Cho (trimethylamine-choline), of tongue tissue between healthy subjects and in patients with squamous cell carcinoma of the tongue, before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patients from the maxillofacial surgery department of the Amiens-Picardie University Hospital treated for histologically confirmed squamous cell carcinoma of the tongue
* Patients who have not yet been treated, either surgically or by neoadjuvant treatment
* Patients with a tumor of minimum dimensions of 15 mm in long axis
* Patients without contraindication to MRI
* Patients over 18 years old
* Patients who have provided free and informed written consent
* Patients benefiting from a social security system

Healthy volunteers:

* Subjects without a history of cancer of the upper aerodigestive tract
* Subjects without contraindication to MRI
* Subjects over 18 years old
* Subjects who have provided free and informed written consent
* Subjects benefiting from a social security system

Exclusion Criteria:

* Patients:
* Patients with a lingual tumor measuring less than 15 mm in long axis

Patients and healthy volunteers:

* Patients with other histological types of cancer, or other locations
* Subjects with a contraindication to MRI
* Subjects under 18 years old
* Pregnant or breastfeeding women
* Persons under guardianship, curators, protection of justice or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
variation in the metabolite TMA-Cho (trimethylamine-choline), between healthy subjects and patients before surgery | day 1
variation in the metabolite TMA-Cho (trimethylamine-choline), between healthy subjects and patients after surgery | day 1

SECONDARY OUTCOMES:
The variation of lipid contents in the tongue tissue between healthy subjects and patients before surgery | day 1
The variation of lipid contents in the tongue tissue between healthy subjects and patients after surgery | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No